CLINICAL TRIAL: NCT01462721
Title: Post-market Study to Evaluate Post-implant Patency Rates of the External Saphenous Vein Support (eSVS®) Mesh in the Treatment of Saphenous Vein Grafts (SVGs) During Coronary Artery Bypass Grafting (CABG) Versus SVGs Without the eSVS Mesh.
Brief Title: The eSVS® Mesh Randomized Post-Market Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Kips Bay Medical, Inc. (Industry)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-001
Record Dates: First submitted 2011-10-26; First posted 2011-10-31 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Coronary Disease; Heart Diseases; Cardiovascular Diseases; Arteriosclerosis; Arterial Occlusive Diseases; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SVG + eSVS Mesh vs Control SVG (Other): Either the Circumflex Coronary Artery (Cx) or the Right Coronary Artery (RCA) will receive the mesh supported vein graft and the native saphenous vein as second and control graft.
  Interventions: Device: eSVS® Mesh

INTERVENTIONS:
Device: eSVS® Mesh — Patients with multi-vessel coronary artery disease who require saphenous vein graft (SVG) coronary artery bypass graft (CABG) surgery of the Right coronary Artery (RCA) and the Circumflex Artery (Cx) due to atherosclerotic coronary artery disease will serve as their own control. They will be randomized to either an SVG+eSVS Mesh to the RCA and an SVG to the Cx or an SVG to the RCA and an SVG+eSVS Mesh to the Cx.
  Other Names: eSVS Mesh; eMesh; external Saphenous Vein Support Mesh

SUMMARY:
The purpose of this study is to evaluate patency rates of the external Saphenous Vein Support (eSVS) Mesh Saphenous Vein Grafts (SVG) and Control SVG at 3-6 months and 24 months.

DETAILED DESCRIPTION:
The study will enroll up to 200 patients at up to 6 sites. Patients will be enrolled upon meeting entrance criteria, including obtaining written informed consent. Eligible patients must be clinically indicated for coronary artery bypass grafting (CABG) using autologous saphenous vein grafts (SVG). The study is a prospective, randomized, repeated measure controlled trial based on each patient receiving one control SVG and one external Saphenous Vein Support (eSVS) Mesh treated SVG. Each patient will be their own control.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with multi-vessel coronary artery disease
* Requires Saphenous Vein Graft (SVG) Coronary Artery Bypass Graft (CABG) surgery of the Right Coronary Artery (RCA) and the Circumflex Artery (Cx) systems due to atherosclerotic coronary artery disease
* SVGs (eSVS Mesh AND Control) meet size requirements as outlined in eSVS Mesh Instructions for Use
* eSVS Mesh implant procedure can be performed as outlined in the eSVS Mesh Instructions for Use
* Are able to give their informed consent

Exclusion Criteria:

* Not able to give informed consent
* No appropriate target coronary vessels
* SVGs (eSVS Mesh or Control) do not meet size requirements as outlined in eSVS Mesh Instructions for Use
* eSVS Mesh implant procedure cannot be performed as outlined in the eSVS Mesh Instructions for Use
* Inability to tolerate or comply with normal post-surgical drug regimen
* Inability to comply with required follow-up coronary angiography/CT

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Patency of external Saphenous Vein Support (eSVS) Mesh Saphenous Vein Graft (SVG) versus Control SVG | 3-6 Months
  Patency of eSVS Mesh and Control SVGs assessed by spiral CT or angiography at 3-6 months following surgery.
Patency and percent stenosis of the eSVS Mesh and Control Saphenous Vein Grafts | 24 Months
  Patency and percent stenosis of the eSVS Mesh and Control SVGs assessed by angiography at 24 months following surgery
The occurrence of any Major Adverse Cardiac Event (MACE) | 3-6 months post implant
  The occurrence of the MACE composite of death, myocardial infarction (Q wave and non-Q wave), stroke, coronary revascularization (i.e. coronary artery bypass surgery or percutaneous coronary intervention), and at 3 to 6-months postimplant.

CONTACTS AND LOCATIONS:
Overall Officials: Randy LaBounty, Study Director — Kips Bay Medical, Inc.
Locations (1):
- University Hospital of Kiel, Kiel, Germany